CLINICAL TRIAL: NCT04130750
Title: Comparison of pCR Rate After Neadjuvant Chemotherapy Guided by Result of in Vitro Cell Culture Drug Sensitivity or Physician's Choice
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PKUPH10B001
Record Dates: First submitted 2019-10-13; First posted 2019-10-17 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Breast Cancer; Neoadjuvant Chemotherapy; Drug Effect
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- treatment of physician's choice (Active Comparator): Patients in this arm will receive neoadjuvant chemotherapy according physician's choice.
  Interventions: Combination Product: treatment of drug screening
- treatment of drug screening (Experimental): Patients in this arm will receive neoadjuvant chemotherapy according results of drug screening vitro.
  Interventions: Combination Product: treatment of drug screening

INTERVENTIONS:
Combination Product: treatment of drug screening — Patients in experimental group will receive a drug screening in vitro to select sensitive chemotherapy drug. And neoadjuvant chemotherapy will be performed according the results of drug screening.

SUMMARY:
Neoadjuvant chemotherapy is an important treatment for breast cancer patients. Patients with triple negative or Her2 enriched subtype who achieved pCR after neoadjuvant chemotherapy would have longer survival. But the overall pCR rate of breast cancer was about 20%. So, different methods have tried to improve pCR rate.Drug sensitivity screening in vitro for different chemotherapy drugs was a promising method for improving pCR rate. But there was no method could select effective drugs accurately for breast cancer patients until now. This study will explore whether drug screening by culturing breast cancer cells in vitro from breast cancer tissue could improve pCR rate compared with traditional neoadjuvant chemotherapy. Breast cancer patients who were candidates for neoadjuvant chemotherapy will be allocated two group. One group will receive neoadjuvant cheotherapy according physician's choices. Another group will receive neoadjuvant chemotherapy according results of drug sensitivity results by in vitro cell culture. pCR rate will be compared between two groups to explore whether drug sensitivity screening could improve pCR rate.

DETAILED DESCRIPTION:
Neoadjuvant chemotherapy for breast cancer could make unresectable breast cancer be resectable and improve breast conservation rate. Patients with triple negative or Her2 enriched subtype who achieved pCR after neoadjuvant chemotherapy would have better survival. But the overall pCR rate of breast cancer was about 20%. And patients with luminal like subtype were less reactive for neoadjuvant chemotherapy. Improving pCR rate maybe could achieve better survival. So, different methods have tried to improve pCR rate.Drug sensitivity screening in vitro for different chemotherapy drugs was a promising method for improving pCR rate. But there was no method could select effective drugs accurately until now. This study will explore whether drug screening by culturing breast cancer cells in vitro from breast cancer tissue could improve pCR rate compared with neoadjuvant chemotherapy depend on physician's choice. 200 breast cancer patients who were candidates for neoadjuvant chemotherapy will be allocated to two group. One group with 100 patients will receive neoadjuvant cheotherapy according physician's choices. Another group with 100 patients will receive neoadjuvant chemotherapy according results of drug sensitivity results by in vitro cell culture. pCR rate will be compared between two groups to explore whether drug sensitivity screening could improve pCR rate.

ELIGIBILITY:
Inclusion Criteria:

* invasive breast cancer candidate for neoadjuvant chemotherapy normal liver and renal function agreed to participate in this experiment

Exclusion Criteria:

* inflammatory breast cancer patients can not receive operation after neoadjuvant chemotherapy distant metastasis

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
pCR rate of neoadjuvant chemotherapy | through study completion, an average of 2 years
  compare which group would have higher pCR rate

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People'S Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No